CLINICAL TRIAL: NCT06091917
Title: Modulating Early-life Nutrition for Childhood Obesity Prevention
Acronym: NutrOb
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PIC-73-23
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Infant Growth; Childhood Overweight
Keywords: Betaine; infant formula; childhood obesity risk; infant growth; one-carbon metabolism
MeSH Terms: conditions — Pediatric Obesity | interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Use of unmodified infant formula for 12 weeks
  Interventions: Dietary Supplement: Regular infant formula
- Betaine supplementation group (Experimental): Use of infant formula supplemented with betaine (final concentration of 100 µmol/L) for 12 weeks
  Interventions: Dietary Supplement: Betaine supplementation in infant formula

INTERVENTIONS:
Dietary Supplement: Betaine supplementation in infant formula — Infant formula will be supplemented with betaine to provide a final concentration of 100 µmol/L in the reconstituted milk. The intervention will last for 12 weeks.
  Arms: Betaine supplementation group
Dietary Supplement: Regular infant formula — Regular (unmodified) infant formula . The intervention will last for 12 weeks.
  Arms: Control group

SUMMARY:
In this study, betaine intake will be increased in formula-fed infants through formula milk supplementation. To do this, a double-blind randomized study has been designed with the supplementation group (infant formula supplemented with betaine) and control group (unsupplemented infant formula). The main objectives of the study are to determine the safety of supplementation and to assess whether there are changes in infant growth.

DETAILED DESCRIPTION:
Childhood obesity is one of the main public health concerns worldwide. Previous results have linked a nutrient called betaine (trimethylglycine) to the risk of childhood obesity. Betaine is a modified amino acid with osmotic properties that participates in the methionine cycle as a methyl group donor. Specifically, previous data demonstrate a link between breast milk betaine content, postnatal growth, and long-term metabolic health, suggesting that betaine supplementation may be an effective strategy for regulating growth trajectories and preventing childhood obesity. This study will assess the effects of increasing betaine intake in formula-fed infants through formula milk supplementation. To do this, a double-blind randomized study has been designed where participants will be randomly assigned to the control group or the supplementation group. The main objectives of the study are to determine the safety of supplementation and to assess whether there are changes in infant growth. Additionally, potential changes in the intestinal microbiome induced by the increase in betaine intake will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age between 17 and 42 years
* Maternal pre-pregnancy BMI equal or higher than 25
* Gestational age at birth > 37 weeks
* No exclusive breastfeeding at time of recruitment

Exclusion Criteria:

* Presence of disease or malformations in the infant
* Infant birth weight < -1 SD (standard deviations)
* Multiple pregnancy
* Elective c-section

Ages: 0 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in weight-for-length z score | From start to the end of treatment at 12 weeks and at 12 months of follow-up
  Weight and length will be measured at different time-points and combined to calculate weight-for-length z scores.
Changes in fecal microbiota composition | At 4 weeks and 12 weeks end of treatment, and at 12 months of follow-up
  Differences in features associated with a healthy mucosal layer and metabolic state (e.g. Bifidobacteria and Akkermansia relative amount). Stool samples will be processed to isolate the bacterial DNA. Microbiome composition will be determined by DNA sequencing.

SECONDARY OUTCOMES:
Infant body composition | At 12 months of follow-up
  Total body and abdominal fat mass measured by dual energy x-ray absorptiometry (DXA) scan
Urine one-carbon metabolite concentration | At 4 weeks and 12 weeks after start of treatment
  Urine samples will be analyzed to quantify betaine content as well as related metabolites (including dimethylglycine, the product of the betaine demethylation reaction

OTHER OUTCOMES:
Infant's DNA methylome | At the end of the 12-week treatment
  DNA will be extracted from infant saliva samples. The DNA methylome will be obtained with array technology.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Joan de Déu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No